CLINICAL TRIAL: NCT01471002
Title: Prospective Study to Evaluate the Efficacy of Percutaneous Cryoablation for Renal Tumours < 4cm in Patients Who Are Not Candidates for Partial Nephrectomy
Brief Title: Study to Evaluate the Efficacy of Percutaneous Cryoablation for Renal Tumours < 4cm in Patients Who Are Not Candidates for Partial Nephrectomy
Acronym: CRYOREIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5062
Record Dates: First submitted 2011-11-03; First posted 2011-11-11 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Renal Tumors Less Than 4 cm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal cancer without nephrectomy (Experimental): patients with renal cancer that cannot be offered a partial nephrectomy
  Interventions: Device: Galil Medical patented 17G Cryoablation Needles

INTERVENTIONS:
Device: Galil Medical patented 17G Cryoablation Needles

SUMMARY:
The main objective is to evaluate the oncologic efficacy of percutaneous cryoablation of renal tumors smaller than 4 cm in patients with renal cancer that cannot be offered a partial nephrectomy. The oncologic outcome will be assessed by the presence or absence of residue or recurrence during a follow-up by MRI performed the first 12 months (M1, M3, M6, M12).

ELIGIBILITY:
Inclusion Criteria:

Patients should have the following characteristics:

* About 75 years, or
* Whatever the age:

  * A context of family-type tumor (VHL, hereditary carcinoma, tubulo-papillary ...);
  * or solitary kidney, when the tumor is not easily accessible for nephron-sparing surgery: Malignant centro-hilar or intra-parenchymal;
  * or in a local recurrence (single or multiple) after partial nephrectomy (within a limit of 3 tumors to be treated);
  * or in a subject with impaired renal function and therefore at risk of severe renal insufficiency (risk defined by a creatinine clearance below 30 ml / min by MDRD formula);
  * and who do not present any contra-indication for cryoablation treatment.

The tumor(s) should meet the following criteria:

* Presence of one to three solid tumors of the native renal parenchyma with a largest diameter less than (or equal to) 40 mm, which corresponds to a maximum volume of about 32 cc, as measured by MRI.
* A preoperative MRI is essential since this technique presents a higher sensitivity. This control will also give more consistency to the evaluation of the radiological semiology at follow-up.
* And its/their location(s) will be accessible to a percutaneous approach.

The search of metastases, including a thoracic CT scan, should be negative.

Exclusion Criter ia:

* - Partial nephrectomy feasible in good technical and oncologic conditions in patients under 75 years and in the absence of family tumors.
* Contraindication to any form of sedation.
* Irreversible coagulopathy
* Tumor> 4cm
* Contraindication to MRI or gadolinium (proven allergy). NB: Patients with a glomerular filtration rate below 30 ml/min/1, 73 m2 will be injected with a single dose of the macrocyclic gadolinium with the highest thermodynamic stability (Dotarem or Prohance), given the united recommendations of AFSSAPS and EMA (European Medicines Agency) [45]. On the contrary, the linear molecules of gadolinium, due to their lower stability, will be contra-indicated because of the risk of systemic nephrogenic fibrosis (FNS).
* Recurrence on the same location after a procedure performed out of the thermoablation protocol.
* Biopsy proven benign tumor
* Predominantly cystic tumor, defined by a necrotic content constituting over one third of tumor volume
* Presence of endo-venous extension, of proven secondary extensions, visceral or in the lymph nodes (especially lung). In this regard, a thoracic CT scan will be routinely required before treatment, according to the recommendations of urological societies.
* Psychiatric disorders and adults under guardianship
* Pregnancy or breastfeeding
* Minor patients
* Legal safeguard
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Suspicious contrast enhancement and progression in size of the cryolesion detected by MRI | 1 year
  The success of cryoablation will be declared if the control at 1 year shows no suspicious contrast enhancement (the suspicious character is defined by significant contrast uptake (>15%) and heterogeneous or nodular or crescent-shape contrast enhancement) and if the cryolesion is not progressing in size compared to early post-ablation control (M1).

CONTACTS AND LOCATIONS:
Overall Officials: Afshin GANGI, PU-PH, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Nouvel Hôpital Civil, Strasbourg, Alsace, France